CLINICAL TRIAL: NCT02528994
Title: A Pilot Study to Test the Effect of Short Term Dietary Serine Supplementation on Circulating Serine Levels
Brief Title: Short Term Dietary Serine Supplementation and Circulating Serine Levels
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI will be leaving the institution and not continuing the study
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Geoffrey Walford, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014D001170
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Serine
Keywords: Dietary supplements; Metabolism
MeSH Terms: interventions — Serine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Serine 6g daily (Experimental): Randomized participants will take 6g daily of dietary serine supplement
  Interventions: Dietary Supplement: L-serine
- Serine 12g daily (Experimental): Randomized participants will take 12g daily of dietary serine supplement
  Interventions: Dietary Supplement: L-serine
- Serine 24g daily (Experimental): Randomized participants will take 24g daily of dietary serine supplement
  Interventions: Dietary Supplement: L-serine
- Serine 48g daily (Experimental): Randomized participants will take 48g daily of dietary serine supplement
  Interventions: Dietary Supplement: L-serine

INTERVENTIONS:
Dietary Supplement: L-serine — Participants will take dietary serine supplementation daily

SUMMARY:
This study will test the effect of short-term, high-dose dietary serine supplementation on circulating levels of serine. Individuals with risk factors for type 2 diabetes will be recruited into the 2 week study. Effects of dietary serine supplementation on glycemic measures will also be explored.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, nutritional intervention study in adults. Subjects will have three visits to the Massachusetts General Hospital Clinical Research Center (CRC) during the 2 week study.

At the first study visit (Visit 1), the following will occur: informed consent; medical and nutritional history assessment; blood pressure, weight and height, fasting blood draw and blood work during a 2 hr oral glucose tolerance test; explanation and instructions for completion of a 4-day food log; randomized assignment to dose of dietary serine supplementation (6g, 12g, 24g, or 48g); provide 7 days of dietary serine supplements; take first dose of supplement with snack; schedule Visit 2 and Visit 3.

Between Visit 1 and Visit 2, participants will complete the Food Log and take the assigned dose of dietary serine supplementation 3 times daily.

Visit 2 will occur 7 days after Visit 1. Subjects will not take dietary serine supplementation prior to Visit 2 activities. At Visit 2, the following will occur: weight and blood pressure; fasting blood draw; administration of assigned dose of dietary serine supplementation with snack after blood work; review of the 4-day food log; provide 7 days of dietary serine supplements completion of anonymous survey to assess tolerability of supplement. Participants will continue to take the assigned dose of dietary serine supplementation 3 times daily between Visit 2 and Visit 3.

Visit 3 will occur 7 days after Visit 2. At Visit 3, the following will occur: weight and blood pressure; review of the 4-day food log; fasting blood draw and blood work during a 2 hr oral glucose tolerance test; completion of study survey to assess tolerability of the supplement.

ELIGIBILITY:
Inclusion Criteria:

* risk factors for type 2 diabetes

Exclusion Criteria:

* known type 2 diabetes
* women who are pregnant, nursing, or not using contraception or abstinence
* taking amino acid supplements during the study or at any time 1 month prior to enrollment in the study
* conditions causing intestinal malabsorption, including celiac disease or a history of intestinal or gastric bypass surgery
* known active liver disease
* currently taking or intending to take during the study duration any medication known to affect glycemic parameters, such as glucocorticoids, growth hormone, or fluoroquinolones
* participation in any other interventional study during the study duration
* inability to adhere to study protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Circulating serine levels | 14 days
  We will measure circulating serine levels after 14 days of intervention

SECONDARY OUTCOMES:
Supplement tolerability | 14 days
  We will assess tolerability of dietary serine supplements after 14 days of intervention
Fasting and post-prandial glucose | 14 days
  We will assess fasting and post-prandial glucose after 14 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Walford, MD, Principal Investigator — Massachusetts General Hospital